CLINICAL TRIAL: NCT07327125
Title: Effect of Skin Closure Techniques on Body Image and Mood in Gynecologic Oncology Patients
Brief Title: Effect of Skin Closure Techniques on Body Image in Women Undergoing Gynecologic Surgery
Acronym: BISGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Mahmut Yassa, Principal Investigator - Gynecologic Oncology Specialist, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCSSH-JINONK-01
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancers; Surgical Wound Closure Techniques; Body Image
Keywords: surgical staples; Subcuticular Sutures; Gynecologic Oncology; Skin Closure Techniques; Body Image; Surgical Wound; Laparotomy; Cicatrix; Anxiety; Depression; Midline Incision; Wound Dehiscence; Wound Complications; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound; Cicatrix; Anxiety Disorders; Depression; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group study. Participants are stratified based on Body Mass Index (<30 vs. ≥30 kg/m²), incision length (<15 cm vs. ≥15 cm), and intra-operative frozen section pathology result (Benign vs. Malignant). Randomization is performed intra-operatively, immediately after the frozen section result is available.
  Allocation uses a 1:1 ratio with permuted blocks of variable sizes (4, 6, 8) to ensure balanced assignment within each stratum. The randomization sequence was pre-generated using a fixed random seed (offline Excel file). Allocation concealment is maintained; the operating surgeon is blinded to future assignments and accesses the next allocation only after the patient is fully eligible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcuticular Suture Group (Experimental): Patients in this group will undergo skin closure using a continuous subcuticular suture technique with absorbable suture material.
  Interventions: Procedure: Continuous Subcuticular Suture
- Interrupted Closure Group (Active Comparator): Patients in this group will undergo skin closure using interrupted techniques. The incision will be closed with either surgical staples (metal clips) or interrupted mattress sutures, depending on the standard practice.
  Interventions: Procedure: Interrupted Skin Closure

INTERVENTIONS:
Procedure: Continuous Subcuticular Suture — Surgical skin closure performed using a continuous technique with absorbable suture material.
  Arms: Subcuticular Suture Group
Procedure: Interrupted Skin Closure — Surgical skin closure performed using interrupted techniques, specifically metal staples or interrupted mattress sutures.
  Arms: Interrupted Closure Group

SUMMARY:
This randomized clinical trial investigates the impact of two different skin closure techniques on body image and mood in women undergoing surgery for gynecologic cancers.

Patients undergoing elective surgery with a midline abdominal incision will be randomly assigned to one of two groups: 1. Interrupted Closure Group: The surgical incision is closed using either metal clips (staples) or separate mattress sutures (individual stitches). 2. Subcuticular Sutures Group: The surgical incision is closed using continuous stitches placed under the skin surface (aesthetic stitching).

The main goal of the study is to determine whether the method of wound closure affects a patient's perception of their body image, cosmetic satisfaction, and levels of anxiety or depression.

Additionally, the study aims to prove that the subcuticular suture technique is safe and does not increase the risk of wound complications (such as infection or wound separation) compared to the other method.

Participants will be asked to complete questionnaires before surgery, and again at 1, 3 and 6 months after surgery to track changes in their feelings and satisfaction with the scar.

DETAILED DESCRIPTION:
Midline abdominal incisions are common in gynecologic oncology, yet the optimal skin closure technique to minimize scar-related psychological distress remains unclear. While staples offer speed, subcuticular sutures may provide superior cosmetic results. This study aims to fill the gap in the literature regarding the specific impact of these closure methods on body image and patient-reported outcomes in gynecologic cancer patients, beyond standard wound complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 years or older.
* Patients scheduled for elective open gynecologic surgery for suspected or confirmed gynecologic malignancy.
* Surgery planned to be performed via a vertical midline laparotomy incision.
* Literate patients capable of reading, understanding, and completing the Body Image Scale (BIS) and Hospital Anxiety and Depression Scale (HADS).
* Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

* History of prior radiotherapy to the abdominal or pelvic region.
* Patients currently receiving chronic immunosuppressive therapy.
* Body Mass Index (BMI) less than 18 kg/m^2 or greater than 40 kg/m^2.
* Presence of cognitive impairment, dementia, or Alzheimer's disease.
* Major psychiatric disorders that prevent the patient from understanding or completing the questionnaires.
* Patients undergoing emergency surgery.

Ages: 17 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Body Image Scale (BIS) Score | Baseline (pre-operative), Post-operative Month 1, Post-operative Month 3 and Post-operative Month 6.
  The Body Image Scale (BIS) is a 10-item questionnaire designed to assess body image changes in cancer patients. Each item is scored on a 4-point Likert scale ranging from 0 (not at all) to 3 (very much). The total score ranges from 0 to 30. Higher scores indicate higher levels of body image distress and dissatisfaction.

SECONDARY OUTCOMES:
Incidence of Wound Complications | Post-operative Month 1, Month 3 and Month 6
  Evaluation of surgical site complications including superficial or deep surgical site infection (SSI), wound dehiscence (separation of wound edges), seroma, and hematoma. Diagnosis is based on clinical examination and standard CDC criteria.
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) Score | Baseline (Pre-operative), Post-operative Month 1, Month 3 and Month 6.
  The HADS is a 14-item self-report screening scale. It consists of two subscales: Anxiety (HADS-A, 7 items) and Depression (HADS-D, 7 items). Each item is scored from 0 to 3. The maximum score for each subscale is 21. Higher scores indicate higher levels of anxiety or depression (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Bora Taşpınar, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the article (text, tables, and figures) will be shared. This includes the data on body image scores, anxiety/depression scores, and wound complications. Data will be available beginning 6 months and ending 5 years following article publication to researchers who provide a methodologically sound proposal. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal approved by an independent review committee or the Principal Investigator. Data will be shared for the purpose of achieving the aims in the approved proposal.